CLINICAL TRIAL: NCT05885360
Title: Istradefylline Effect on Parkinson's Disease Tremor, Motor Symptoms and Non-motor Symptoms
Brief Title: Istradefylline Effect Protocol on Parkinson's Disease Tremor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005472
Record Dates: First submitted 2023-02-07; First posted 2023-06-01 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease; Tremor
MeSH Terms: conditions — Parkinson Disease; Tremor | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Istradefylline 20 and 40 mg (Experimental): The study intervention will be to add 20 mg Istradefylline for 2 weeks, following which the dose will be increased to 40 mg daily for the remainder of the 24 weeks.
  Interventions: Drug: Istradefylline Pill

INTERVENTIONS:
Drug: Istradefylline Pill — Istradefylline targets adenosine A2A receptors in the basal ganglia, by inhibiting the indirect pathway It is an adjunctive treatment to carbidopa-levodopa indicated to improve "on" time and decrease off time.
  Other Names: NOURIANZ

SUMMARY:
This is an investigator-initiated trial. In this 6-month open label, single arm, exploratory pilot study, the investigator intends to enroll a pilot sample of 25 patients with Parkinson's disease who are being started on the novel FDA approved medication "Istradefylline'' as an add on therapy for management of their motor symptoms (based on the judgment of the movement disorders specialist, if patients are in sub-optimal management of their symptoms on maximum tolerable dose of their dopaminergic medications). The investigator will evaluate their motor symptoms before starting the new medication, including their MDS-UPDRS total and MDS-UPDRS-III scores.

DETAILED DESCRIPTION:
In this 6-month open label, single arm, exploratory pilot study, the investigator intends to enroll a pilot sample of 25 patients with Parkinson's disease who are being started on the novel FDA approved medication "Istradefylline'' as an add on therapy for management of their motor symptoms (based on the judgment of the movement disorders specialist, if patients are in suboptimal management of their symptoms on maximum tolerable dose of their dopaminergic medications). The investigator will evaluate their motor symptoms before starting the new medication, including their MDS-UPDRS total and MDS-UPDRS-III scores.

Based on data from an early experience limited data set within our clinical practice of patients taking Istradefylline, the investigator noted improvement in motor symptoms on PDRS-III. The investigator evaluated the degree of tremor with a tremor quantifying software before and after 8 weeks of therapy. Tremor amplitude, frequency and severity improved in the first two patients based on said parameters.

Secondary analysis in week 24 will include all aforementioned assessments. The investigator will compare their score and results before and after the medication.

The therapeutic intervention will consist of evaluating the effect of the addition of Istradefylline 40 mg daily (after two weeks of Istradefylline 20 mg daily) in patients already on levodopa and other anti- parkinsonian treatments. Patients will be screened based on inclusion and exclusion criteria. Enrolled patients will need to be on a stable regimen of all their concomitant medications for at least 30 days prior to baseline visit. All PD concomitant medications are allowable. Participants must also have a MOCA (Montreal Cognitive Assessment) of 22 or greater, and the absence of a diagnosis of dementia.

Tremor score will be clinically defined by the presence of a sum score of at least 8 of 32 of the MDS-UPDRS tremor items 16, 20, and 21 (referred to as tremor score). The generation of this sum score is based on the validity of the MDS-UPDRS regarding tremor, 19 and the clinical experience, that the MDS-UPDRS tremor items reflect different but similarly important aspects of Parkinsonian tremor, including the impairment of activities of daily living by tremor.

ELIGIBILITY:
Inclusion Criteria:

* · Written informed consent

  * Capable of providing informed consent and complying with study procedures
  * Clinical diagnosis of Parkinson's disease according to the United Kingdom Brain Bank criteria which includes the following.
  * Bradykinesia
  * At least one of the following:
  * Muscular righty
  * 4-6 Hz rest tremor
  * Postural instability not caused by primary visual, vestibular, cerebellar, or proprioceptive dysfunction
  * Must be on a stable regimen of all current concomitant medication, including carbidopa-levodopa for at least 30 days prior to baseline visit
  * Participants also have a MOCA (Montreal Cognitive Assessment) score of 22 or greater
  * Study subjects are willing to present for all study visits and take medication.
  * The MDS-UPDRS I-III will be used to assess a baseline tremor score

Exclusion Criteria:

* · Diagnosis of dementia - defined by NIH as the loss of cognitive functioning such as thinking, remembering, and reasoning, to such an extent that it interferes with a person's daily life and activities.

  * Parkinson's plus syndromes or any other disorder other than idiopathic Parkinson's disease
  * Moderate to severe dyskinesia is defined as:
  * Moderate: Dyskinesias impact on activity to the point that the patient usually does not perform some activities or does not usually participate in some social activities during dyskinetic episodes
  * Severe: Dyskinesia impacts activities to the point that the patient usually does not perform most activities or participate in most social activities during dyskinetic episodes
  * Patients with severe cardiac disease or congestive heart failure
  * Severe uncontrolled orthostatic hypotension
  * Psychosis or psychotic symptoms that would raise concern for safe use of IST, as indicated by domains A (delusions) and B (hallucinations) of the Neuropsychiatric Inventory (NPI), and defined as a score of ≥ 4 on either the A (frequency x severity) or B (frequency x severity) scales of the NPI
  * Active neoplastic disorder
  * Current treatment with strong CYP3A4 inhibitors
  * Current treatment with strong CYP3A4 inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
To observe the effect of Istradefylline on tremor in PD patients. | 8 weeks
  · Evaluation of changes in MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) III tremor score
  ·· Evaluation of changes in the Movement Disorders Society - United Parkinson's Disease Rating Scale part III tremor score, with the minimum value being 0 and the maximum value being 4 for each sub-scale (rest, kinetic and postural), with a higher score signifying a worse outcome.

SECONDARY OUTCOMES:
To evaluate the changes in MDS-UPDRS part I (non-motor) in PD patients with tremor. | 24 weeks
  * Evaluation of changes in MDS-UPDRS part I (non-motor)
  * Evaluation of changes in Movement Disorders Society- United Parkinson's Disease Rating Scale Part I (non-motor) with a minimum score being 0 and a maximum score being 52, where a higher score signifies a worse outcome
To evaluate the changes in MDS-UPDRS II motor symptoms in PD patients with tremor. | 24 weeks
  * Evaluation of changes in MDS-UPDRS II motor experiences of daily living (MEDL) score
  * Evaluation of changes in Movement Disorders Society- United Parkinson's Disease Rating Scale Part II motor experiences of daily living (MEDL) score with a minimum score of 0 and a maximum score of 52 with a higher score signifying a worse outcome.
To evaluate the changes in cognition, mood and behavior in Parkinson's disease patients treated with Istradefylline. | 24 weeks
  * Evaluation of changes in EQ5D
  * To evaluate the changes in cognition, mood and behavior in Parkinson's disease patients treated with Istradefylline by evaluating the change in score in the EuroQol 5 Dimension 5 Level (EQ5D), with a minimum score of 1 and a maximum score of 15, with a higher value being associated with a worse outcome.
To evaluate the the Geriatric depression scale (GDS) in PD patients with tremor. | 24 weeks
  - To evaluate the changes in cognition, mood and behavior in Parkinson's disease patients treated with Istradefylline by evaluating the change in score in the Geriatric depression scale (GDS), with a minimum score of 0 and a maximum score of 10, where a higher score signifies a worse outcome.
To evaluate the effect of Istradefylline on activities of daily living in PD patients with tremor. | 24 weeks
  - To evaluate changes due to adjustments to individual concomitant medications in response to adverse events due to Istradefylline and changes in the Movement Disorders Society- United Parkinson's Disease Rating Scale Part III tremor score.
To assess the utility of a tremor capturing application such as Mindsquare app. | 24 weeks
  - To assess the utility of a tremor capturing application (Mind-square) to measure tremor severity (amplitude as measured by the average displacement in the Z axis)
To assess changes in motor impairment using the Right Eye eye- tracking technology. | 24 weeks
  - To assess changes in motor impairment using the Dynamic Vision test, a part of the Right Eye eye-tracking technology, to measure changes in pursuits, fixations and saccades eye movements, which a minimum score of 0 percentile and a maximum score of 100th percentile, with the higher score signifying a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Pagan, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, McLean, Virginia, United States

IPD SHARING:
Plan to Share IPD: No